CLINICAL TRIAL: NCT02512198
Title: Electronic Prescription Data to Improve Primary Care Prescribing
Acronym: EPIPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UREC15066
Record Dates: First submitted 2015-07-23; First posted 2015-07-30 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Physician's Practice Patterns
Keywords: Professional Practice; General Practitioners; Inappropriate Prescribing; Persuasive Communication; Information Theory; Feedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bronchodilators (Experimental): Prescription Data Feedback to GP Practices - practices will be fed back data for people with presumed asthma who have either been dispensed more than 12 short-acting beta-agonist bronchodilators in the last 12 months who are not concurrently prescribed inhaled corticosteroids (poor asthma control with inadequate prevention) or been dispensed a long-acting beta-agonist bronchodilator as a single agent in the last 12 months who are not or are only infrequently concurrently prescribed inhaled corticosteroids (potentially harmful prescribing). To minimise inclusion of people with COPD, patient aged 35 years and older prescribed long-acting antimuscarinic bronchodilators will be excluded.
  Practices in the bronchodilator arm are controls for the antibiotic experimental arm (below).
  Interventions: Behavioral: Prescription Data Feedback to GP Practices
- Antibiotics (Experimental): Prescription Data Feedback to GP Practices - number of women in the GP practice aged 12 years and older dispensed more than 6 courses of urinary tract infection (UTI) antibiotics in the last year. UTI antibiotics are defined as trimethoprim, nitrofurantoin, co-trimoxazole, quinolones and cefalexin.
  Practices in the antibiotic arm are controls for the bronchodilator experimental arm (above).
  Interventions: Behavioral: Prescription Data Feedback to GP Practices

INTERVENTIONS:
Behavioral: Prescription Data Feedback to GP Practices — GP practices will be randomly assigned to receive reports on one of the two topics. They will get these three times at six-monthly intervals. Within the feedback, alongside the patient-level analysis, there will be action-orientated messages to guide the GP practice.

SUMMARY:
This is a randomised controlled study to evaluate the effect of providing prescribing feedback that includes individual patient data to General Practitioners (GP) in Scotland on high risk or low quality prescribing.

DETAILED DESCRIPTION:
This study makes use of data held in the Prescription Information System (PIS), the national database available to national health service (NHS) health boards in Scotland, on all prescriptions dispensed by community pharmacists which include the unique patient identifier for Scotland (CHI).

The design is a two parallel arm cluster randomised trial with general practices as the unit of randomisation to whom the feedback intervention is directed, and outcomes measured at patient level. Both arms receive the same active interventions but focused on different topics, with each acting as control to the other.

The primary outcome in the asthma arm is a composite of measure of potentially high-risk asthma prescribing (multiple short acting beta-agonists or single agent long acting beta-agonists both in the absence of inhaled corticosteroid therapy).

The primary outcome in the urinary tract infection antibiotic arm is a measure of repeated use of single (likely long-term prevention) or multiple (repeated treatment courses) urinary tract infection antibiotics.

Within the feedback, alongside the patient-level analysis, there will be action-orientated messages to guide the GP practice.

GP practices will get the reports three times at six-monthly intervals.

ELIGIBILITY:
Inclusion Criteria:

* GP practices in the participating Health Board area (NHS Greater Glasgow and Clyde)

Exclusion Criteria:

* GP practices with registered list sizes <250 patients (all of these are unusual practices in various ways, for example serving the homeless or people with challenging behaviour).
* GP practices with <80% of prescriptions for inhaled bronchodilators and UTI antibiotics in the prescription database with a recorded patient identifier for each month from January 2014 to December 2014.
* GP practices which were created after 1 January 2015.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2015-07; Primary Completion 2017-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Number of people identified by the measures of high risk or low quality prescribing | 12 months

SECONDARY OUTCOMES:
Cost-effectiveness of feedback | 12 months
  The economic evaluation will estimate costs and benefits using the cost perspective of the NHS, it will take account medicines cost, costs within the GP practice and use of other NHS services.

CONTACTS AND LOCATIONS:
Overall Officials: Sean PD MacBride-Stewart, MSc, Principal Investigator — University of Dundee
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom